CLINICAL TRIAL: NCT04114253
Title: Evaluation of the Clinical Performance of the Quantra System With the QStat Cartridge in Liver Transplant
Brief Title: QStat in Liver Transplant
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-029
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Blood Loss, Surgical
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Liver transplant patients: Adult patients undergoing deceased donor liver transplantation.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra QStat Cartridge

SUMMARY:
This study will assess the clinical performance of the Quantra System with the QStat Cartridge in the liver transplant population.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic propoerties of a whole blood sample during coagulation. The Quantra QStat Cartridge was developed to monitor hemostasis in the trauma and liver transplant populations which may experience a range of coagulopathies of various etiologies including fibrinolytic defects.

This single-center, prospective, observational stuey will evaluate the performance of the Quantra System with the QStat Cartridge as compared to corresponding measures determined using the TEG 5000.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is undergoing deceased donor liver transplant and is a candidate for a TEG test to be performed to access coagulopathy during surgery.
* Subject is willing to participate, and is willing to consent (either prospectively or by deferred consent)

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is known to have received antifibrinolytic therapy immediately prior to the start of liver transplantation surgery.
* Subject is unable to provide written informed consent (either prior to performing any study related procedures or by deferred consent)
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects 18 years or older undergoing deceased donor liver transplant.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time results to TEG R results | Baseline, after induction of anesthesia, before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | Baseline, after induction of anesthesia, before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Lysis results to TEG LI30 results | Baseline, after induction of anesthesia, before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Time results to TEG R results | During surgery
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | During surgery
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Lysis results to TEG LI30 results | During surgery
  Coagulation function assessed by Quantra and TEG 5000

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No